CLINICAL TRIAL: NCT00907192
Title: The Influence of Patients' Knowledge, Attitudes and Beliefs on Self Reported Deviations From Opioid Analgesic Prescription: an Exploratory Survey
Brief Title: Self Reported Deviations From Opioid Analgesic Prescription
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0019
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Advanced Cancers
Keywords: Cancer; Opioid analgesic prescriptions; Narcotic pain drugs; Self-report; Questionnaire; Interview; Actual use; Doctor-prescribed use; Frequency of deviation
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Opioids: Personal Interview and Questionnaire of Advanced cancer patients, taking narcotic pain drugs (opioids).
  Interventions: Behavioral: Personal Interview; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Personal Interview — Interview questions about use of pain drugs and other knowledge and/or attitudes about them. Take about 5-10 minutes to complete.
Behavioral: Questionnaire — 5 short questionnaires about use of pain drugs, attitudes about the pain drugs and their use, and concerns about use of these pain drugs. Take about 10-15 minutes to complete.
  Other Names: Survey

SUMMARY:
Primary Objective:

1. To determine the frequency of self-reported over and under use of opioid analgesics in patients with advanced cancer. Patients with advanced cancer are those patients who have been described to have either one of the following: recurrent disease, those that have failed multiple chemotherapies (more than second line therapy), locally advanced disease, and metastatic disease.

Secondary Objectives:

1. To determine the association between patients' knowledge, attitudes and beliefs about opioids, and frequency of deviation in opioid use with patients' demographic information.
2. To determine association between alcohol abuse/chemical coping and self-reported deviations in opioid use.
3. To determine the association between the use of opioids and patient-related barriers to opioid use.

DETAILED DESCRIPTION:
Screening:

Before you start the study, the research nurse will check your medical record to see if you are eligible to take part in this study. Information will be recorded about your demographics (such as age, marital status, ethnicity, education level, and gender), medical history (such as the type of cancer and level of pain), and prescriptions (such as the name of any opioid drugs, doses, and schedule).

Interview Process:

If you are found to be eligible to take part in this study, you will be interviewed by the study staff before a regular visit with your doctor. You will be asked some questions about your use of pain drugs and other knowledge and/or attitudes that you may have about them. You may also be asked for general information (such as your age, marital status, or educational level) if it was not available in your chart and medical record.

Questionnaires:

After the interview, you will complete 5 short questionnaires about your use of pain drugs, your attitudes about the pain drugs and their use, and concerns that you may have about your use of these pain drugs.

It will take about 5-10 minutes for the interview and another 10-15 minutes to complete all the questionnaires.

Your interview and questionnaire responses will not be shared with your regular doctor unless the study staff feels that you maybe be at harm. If you feel you need a doctor's opinion about anything that is asked in the interview and/or questionnaires, please contact your doctor.

Confidentiality:

Your interview and questionnaire responses will only be used for this research study and will not be shared with your family members.

Length of Study:

After completing the interview and questionnaires, your participation in this study will be over.

This is an investigational study. Up to 200 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years old and have a diagnosis of advanced cancer.
2. Patients must be given prescriptions for around the clock (ATC) and as needed (for breakthrough pain) oral opioids for cancer pain on the previous visit to the Palliative Care Clinic.
3. Patients must be able to understand, read, write, and speak English.
4. Patients must have no clinical evidence of cognitive impairment, as determined by the primary palliative care physician.
5. Patients must sign an informed consent.

Exclusion Criteria:

1. Patients who have the caregiver as the primary person that does the management of opioid medication intake will be excluded as analysis is focused on patients' and not the family or caregivers' knowledge, attitudes and beliefs as it relates to the primary objective.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients least 18 years old, diagnosised advanced cancer, and are taking narcotic pain drugs (opioids).
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of Persons with Advanced Cancer who Self-report Opioid Analgesics Over/Under | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org